CLINICAL TRIAL: NCT00694954
Title: A Randomized Controlled Trial of Capsule Endoscopy vs Standard Care in Patients With Iron Deficiency Anemia With Suspected Obscure / Occult Gastrointestinal Bleeding
Brief Title: Capsule Endoscopy vs Standard of Care for Obscure Intestinal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Calgary Health Region (Other)
Responsible Party: Principal Investigator, Dr. Robert Hilsden, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E20270; Internal tracking #1763
Record Dates: First submitted 2007-12-14; First posted 2008-06-11 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; Wireless capsule endoscopy; Obscure-occult gastrointestinal bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Wireless capsule endoscopy
  Interventions: Device: Diagnostic Test - Given Imaging Pillcam
- 2 (Active Comparator): Standard Care
  Interventions: Other: Diagnostics

INTERVENTIONS:
Device: Diagnostic Test - Given Imaging Pillcam — Procedure performed once only after randomization. If procedure is incomplete due to a number of variables, procedure may possibly need to be repeated.
  Diagnostic possibilities: normal exam, active bleeding, potential source of bleeding (angiodysplasia, ulcer, tumor)
  Other Names: Capsule endoscopy; Given Imaging Pillcam; Pill camera
  Arms: 1
Other: Diagnostics — Any other diagnostic tests (if not already performed) that the referring or attending physician deems necessary aside from Wireless Capsule Endoscopy.
  Arms: 2

SUMMARY:
The role of capsule endoscopy (CE) in patients with obscure / occult gastrointestinal (GI) bleeding remains unclear. This pragmatic randomized controlled trial is designed to determine the diagnostic yield and clinical outcomes of patients with obscure GI bleeding who receive CE compared to those who receive usual standard care.

DETAILED DESCRIPTION:
Patients with iron deficiency anemia from suspected occult GI bleeding will be randomized to receive CE or usual standard care following a negative gastroscopy and colonoscopy. Our primary outcome measure (diagnostic yield) and secondary outcome measures (noted below) will be determined after one year of followup. Patients with have a minimum of one year of clinical followup. Direct health care costs in each arm of the study will be determined after a minimum of two years of followup.

An economic evaluation based on the results of the clinical trial is also planned.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age over 18years with iron deficiency anemia (IDA). IDA is defined as hemoglobin <137g/L in men or <120g/L in women with serum ferritin level <22ug/L in men and <10ug/L in women.
2. Eligible patients should have a negative gastroscopy and negative colonoscopy within 1 year prior to entry into study.
3. Negative celiac screen and /or negative small bowel biopsies

Exclusion Criteria:

1. Overt gastrointestinal bleeding
2. Premenopausal women with menorrhagia
3. Known or suspected small bowel obstruction
4. Serious medical co-morbidities precluding surgery given the risk of capsule impaction
5. Pregnancy
6. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-02; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
diagnostic yield | 48 weeks

SECONDARY OUTCOMES:
number of blood transfusions | 48 weeks
number of hospitalizations for GI bleeding/anemia | 48 weeks
number of GI-related procedures and investigations | 48
procedure-related complications | 48
quality of life | 48
  measured by 1) SF36 - 8 domains + PCS/MCS, 2) GI Quality of Life Index (GIQLI), 3) EQ-5D - index + visual analogue scale
health care costs | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Dube, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada